CLINICAL TRIAL: NCT02051296
Title: A Trial of Minocycline for Pain After Carpal Tunnel and Trigger Release
Brief Title: Minocycline to Reduce Pain After Carpal Tunnel Release
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Collaborators: Stanford University (Other)
Responsible Party: Principal Investigator, Catherine Curtin, Staff Physician, VA Palo Alto Health Care System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RX000487
Record Dates: First submitted 2014-01-26; First posted 2014-01-31 (Estimated); Results first posted 2018-06-11 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-05

CONDITIONS: Chronic Pain; Post-operative Pain
MeSH Terms: conditions — Chronic Pain; Pain, Postoperative | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- minocycline (Experimental): perioperative minocycline for 5 days, starting 2 hours prior to surgery then 100mg BID
  Interventions: Drug: Minocycline
- Placebo (Placebo Comparator): PLacebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Minocycline — RCT blinded placebo trial
  Other Names: Minocycline Hydrochloride
  Arms: minocycline
Drug: placebo — RCT blinded placebo trial
  Arms: Placebo

SUMMARY:
The investigators are looking at whether peri-operative minocycline will reduce the duration of pain after minor hand surgery: carpal tunnel release and trigger finger release.

The investigators' hypothesis is that minocycline will reduce post-operative pain.

DETAILED DESCRIPTION:
This is a double blinded randomized controlled trial. Patients are given 100mg of minocycline 2 hours prior to their procedure and then 100mg two times a day for 5 days. The subjects are then contacted daily to check their level of pain. The investigators' outcome of interest is time to pain resolution.

The investigators will perform a futility analysis to assess if a larger trial would be a reasonable next step after this pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Adult, Veteran,

Exclusion Criteria:

* Kidney failure, Liver failure, thrombocytopenia, ALS, SLE, Frailty, unable to understand survery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2012-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Curtin, MD, Principal Investigator — Palo Alto Veterans Hsopital
Locations (1):
- Palo Alto VA, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Minocycline: perioperative minocycline for 5 days, starting 2 hours prior to surgery then 100mg BID for 5 days
  Minocycline: RCT blinded placebo trial
- Placebo: Placebo: two pills 2 hours prior to surgery then 1 pill BID
  placebo
Period: Overall Study
Arm/Group | Minocycline | Placebo
Started | 66 | 65
Received Allocated Intervention | 59 | 58
Completed | 58 | 56
Not Completed | 8 | 9
Not completed — Lost to Follow-up | 1 | 2
Not completed — withdraw prior to treatment | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Minocycline | Placebo | Total
Number analyzed (Participants) | 58 | 56 | 114
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 34 | 71
  >=65 years | 21 | 22 | 43
Age, Continuous [Mean (Full Range); unit: years] | 60 [27 to 76] | 60 [26 to 79] | 60 [26 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 22
  Male | 45 | 47 | 92
Region of Enrollment [Number; unit: participants]
  United States | 58 | 56 | 114
Brief Pain Inventory(Short Form) [Median (Full Range); unit: units on a scale] — The Brief Pain Inventory measures two constructs.
  Each item is rated from 0, no pain/no interference, to 10, pain as bad as you can imagine/worst interference.
  1. Pain severity score:calculated from the 4 items about pain intensity. It is scored as the mean/median of the seven interference items when all 4 items are not missing.
  2. Pain interference score: It is scored as the mean/median of the seven interference items. This median can be used if more than 50%, or four of seven, of the total items have been completed on a given administration.
  units on a scale
    Brief Pain Inventory Severity Score | 5 [0 to 9] | 5 [1 to 10] | 5 [0 to 10]
    Brief Pain Inventory Interference Score | 3 [0 to 9] | 4 [0 to 9] | 3 [0 to 9]
screen for Posttraumatic Stess Symptoms(SPTSS) [Median (Full Range); unit: units on a scale] — The Brief SPTSS is a 17-item self-report measure that assesses DSM-IV symptoms of PTSD. For this survey, the respondents rated items on an 4-point scale ranging from 0 ("not at all") to 4 ("more than once everyday"). The points were sum across all items for each participant.
  A median score of 12 or higher has been used as the cut-off for psychological distress on this scale. [Dr. Eve Carlson personal communication] We dichotomized as low distress with a score less than 16 and high score 16 or greater. the range was from 0 to 68 points.
  units on a scale | 10 [0 to 58] | 9 [0 to 68] | 9 [0 to 68]
Quick Disability Arm Shoulder and Hand(qDASH) [Median (Full Range); unit: units on a scale] — The Quick Disability Arm Shoulder and Hand (QDASH) is a continuous variable to measure upper extremity physical function and disability. The QDASH consists of 11 items from the original 30-item DASH and has similar reliability and correlation with psychological stress as the full DASH. The scores range from 0 (best function) to 100 (worst function).
  units on a scale
    Quick Disability Arm Shoulder and Hand | 35 [5 to 91] | 45 [5 to 91] | 41 [5 to 91]
    Arm Shoulder and Hand Work | 44 [0 to 44] | 44 [0 to 88] | 44 [0 to 100]
    Arm Shoulder and Hand Play | 50 [0 to 100] | 56 [0 to 100] | 50 [0 to 100]
Beck Depression Inventory-II(BDI-II) [Median (Full Range); unit: units on a scale] — Beck Depression Inventory-II (BDI-II) is a widely used validated measure of depressive symptoms. It consists of 21 groups if statements. A score greater than 16 is the cutoff for depression.
  scoring: The sum of the score for each of the 21 questions.
  depression ranges:
  Low 1-10 Normal ups and downs 11-16 Mild mood disturbance Moderate 17-20 Borderline clinical depression 21-30 Moderate depression Significant 31-40 Severe depression Over 40 Extreme depression
  units on a scale | 9 [0 to 39] | 8 [0 to 38] | 8 [0 to 39]
RAND 36 Item Health Survey( short form(SF-36)) [Median (Full Range); unit: units on a scale] — All ques. are scored on a scale from 0(lowest)-100(highest) functioning (50 avg.)
  Scoring: First, recoded per the scoring key. Scores represent the percentage of total possible score achieved. Second, avg. non missing items in same scale to create 8 scale scores .Scores represent the median for all items in the scale that the respondent answered.
  Physical Functioning 10 Items Role Functioning/physical 4 Items Role Functioning/emotional 3 Items Energy/fatigue 4 Items Emotional well-being 5 Items Social functioning 2 Items Pain 2 Items General Health 5 Items Health Change 1 Item
  units on a scale
    Physical Component Score | 57 [42 to 72] | 58 [39 to 73] | 57 [39 to 73]
    Mental Component Score | 48 [35 to 56] | 47 [33 to 62] | 47 [33 to 62]

OUTCOME MEASURES:

1. Primary Outcome: Time to Pain Resolution
Description: the time until patient answers no pain at surgical site for three consecutive days
Time Frame: up to 365 days
Population: 94 CTR enrolled and randomized, 83 completed and reached endpoint (43 in minocycline group and 40 in placebo group) 37 TFR enrolled and randomized, 31 completed and reached endpoint (15 in minocycline group and 16 in placebo group)
Measure: Median (Full Range); unit: DAYS
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 58 | 56
DAYS | 17 [3 to 365] | 15 [3 to 365]

ADVERSE EVENTS:
Time Frame: The patients were followed up for 6 months after surgery.
Arm/Group | Minocycline | Placebo
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/56
Other Adverse Events (participants affected / at risk) | 4/58 | 3/56
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minocycline (N=58) | Placebo (N=56)
dizziness (General disorders) | 4 (5) | 3 (4) — >7/10 by self report

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No